CLINICAL TRIAL: NCT02413437
Title: The Multi-center Study of Percutaneous Focal Liver Lesions Biopsy Guided by Contrast-Enhanced Ultrasound
Brief Title: A Trial on Contrast-enhanced Ultrasound Versus Conventional Ultrasound Guided Biopsy of Liver Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Kun Yan, Beijing Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014YJZ31
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Liver Neoplasms
Keywords: contrast-enhanced ultrasound; biopsy
MeSH Terms: conditions — Liver Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CEUS guided biopsy (Experimental): Biopsy was operated under contrast-enhanced ultrasound-guided
  Interventions: Other: CEUS guided biopsy; Device: Ultrasound
- US guided biopsy (Other): Biopsy was operated under conventional ultrasound-guided
  Interventions: Other: US guided biopsy; Device: Ultrasound

INTERVENTIONS:
Other: CEUS guided biopsy — Biopsy was operated under contrast-enhanced ultrasound-guided.
  Arms: CEUS guided biopsy
Other: US guided biopsy — Biopsy was operated under conventional ultrasound-guided.
  Arms: US guided biopsy
Device: Ultrasound

SUMMARY:
The purpose of this study is to estimate the clinical value of contrast-enhanced ultrasound in percutaneous biopsy for liver occupied lesion.

DETAILED DESCRIPTION:
The patients with liver neoplasms who need receive percutaneous biopsy were randomized into contrast-enhanced ultrasound(CEUS) group and conventional ultrasound(US) group.The aims include:

1. Comparison the diagnostic accuracy rate, specificity and sensitivity between CEUS and US group.
2. Comparison the diagnostic accuracy rate specificity and sensitivity between smaller(<3cm) and larger(≥3cm) nodule group.
3. To explore operating strategy of contrast-enhanced ultrasound guided biopsy.
4. To evaluate economic efficiency of contrast-enhanced ultrasound guided biopsy compared with conventional ultrasound guided biopsy.

ELIGIBILITY:
Inclusion Criteria:

* patients with liver occupied lesion who cannot be diagnosed by imaging examination or need pathological results

Exclusion Criteria:

* severe anemia
* PLT<60000/mm3,prothrombin activityprothrombin time activity<70%
* women during menstruation, pregnancy, child birth and baby nursing period
* patients with severe mental disorder
* cardiopulmonary failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2088 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 12 months
  diagnostic accuracy=（true positive+ ture negative)/number of parcitipants

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yan, master, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Rossi P, Sileri P, Gentileschi P, Sica GS, Forlini A, Stolfi VM, De Majo A, Coscarella G, Canale S, Gaspari AL. Percutaneous liver biopsy using an ultrasound-guided subcostal route. Dig Dis Sci. 2001 Jan;46(1):128-32. doi: 10.1023/a:1005571904713. PMID 11270776
- [Result] Schlottmann K, Klebl F, Zorger N, Feuerbach S, Scholmerich J. Contrast-enhanced ultrasound allows for interventions of hepatic lesions which are invisible on convential B-mode. Z Gastroenterol. 2004 Apr;42(4):303-10. doi: 10.1055/s-2004-812712. PMID 15095120
- [Result] Wu W, Chen MH, Yin SS, Yan K, Fan ZH, Yang W, Dai Y, Huo L, Li JY. The role of contrast-enhanced sonography of focal liver lesions before percutaneous biopsy. AJR Am J Roentgenol. 2006 Sep;187(3):752-61. doi: 10.2214/AJR.05.0535. PMID 16928941
- [Result] Bang N, Bachmann Nielsen M, Vejborg I, Mellon Mogensen A. Clinical report: contrast enhancement of tumor perfusion as a guidance for biopsy. Eur J Ultrasound. 2000 Dec;12(2):159-61. doi: 10.1016/s0929-8266(00)00108-7. PMID 11118924
- [Result] Caturelli E, Biasini E, Bartolucci F, Facciorusso D, Decembrino F, Attino V, Bisceglia M. Diagnosis of hepatocellular carcinoma complicating liver cirrhosis: utility of repeat ultrasound-guided biopsy after unsuccessful first sampling. Cardiovasc Intervent Radiol. 2002 Jul-Aug;25(4):295-9. doi: 10.1007/s00270-001-0123-6. Epub 2002 Mar 27. PMID 12324817
- [Derived] Wu W, Jing X, Xue GQ, Zhu XL, Wang J, Du RQ, Lv B, Wang KF, Yan JP, Zhang ZY, Li MD, Kono Y, Yan K. A Multicenter Randomized Controlled Study of Contrast-enhanced US versus US-guided Biopsy of Focal Liver Lesions. Radiology. 2022 Dec;305(3):721-728. doi: 10.1148/radiol.212317. Epub 2022 Aug 2. PMID 35916680